CLINICAL TRIAL: NCT01174264
Title: Evaluation of Food Effect on Pharmacokinetics of GDC-0449, an Inhibitor of Hedgehog Signaling
Brief Title: Evaluation of Food Effect on Pharmacokinetics of Vismodegib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03099; NCI-2012-03099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 8395; 09-149-B (Other: University of Chicago Comprehensive Cancer Center); 8395 (Other: CTEP); P30CA014599 (NIH); U01CA069852 (NIH)
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — HhAntag691

ARMS (3):
- Arm I (vismodegib on empty stomach) (Experimental): Patients receive a single dose of vismodegib PO on an empty stomach. Beginning 7 days later, patients receive vismodegib PO on an empty stomach daily on days 1-28.
  Interventions: Other: Pharmacological Study; Drug: Vismodegib
- Arm II (vismodegib after high fat meal) (Experimental): Patients receive a single dose of vismodegib PO after eating a high fat meal. Beginning 7 days later, patients receive vismodegib PO on an empty stomach daily on days 1-28.
  Interventions: Other: Pharmacological Study; Drug: Vismodegib
- Arm III (vismodegib after low fat meal) (Experimental): Patients receive a single dose of vismodegib PO after eating a low fat meal. Beginning 7 days later, patients receive vismodegib PO after eating a meal daily on days 1-28.
  Interventions: Other: Pharmacological Study; Drug: Vismodegib

INTERVENTIONS:
Other: Pharmacological Study — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This randomized clinical trial studies the effect of food on the pharmacokinetics of vismodegib. Studying the effects of meals on the absorption of vismodegib may help doctors prescribe correct doses and label the drug accurately.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of prandial states on the pharmacokinetic parameters of GDC-0449 (vismodegib).

II. To evaluate the effect of fat content of meals on the pharmacokinetic parameters of GDC-0449.

SECONDARY OBJECTIVES:

I. To evaluate the effect of prandial states and fat content of meals on the safety profile of GDC-0449.

II. To describe any anticancer activities of GDC-0449.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive a single dose of vismodegib orally (PO) on an empty stomach. Beginning 7 days later, patients receive vismodegib PO on an empty stomach daily on days 1-28.

ARM II: Patients receive a single dose of vismodegib PO after eating a high fat meal. Beginning 7 days later, patients receive vismodegib PO on an empty stomach daily on days 1-28.

ARM III: Patients receive a single dose of vismodegib PO after eating a low fat meal. Beginning 7 days later, patients receive vismodegib PO after eating a meal daily on days 1-28.

In all arms, treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced malignancies (except for leukemias) refractory to standard of care therapy, or for whom no standard of care therapy is available
* Measurable or non-measurable disease
* An anticipated life expectancy > 3 months
* Karnofsky performance status of > 70%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 48 hours prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449

  * Female subjects of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female subjects may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to menopausal (no menstrual period) for 24 consecutive months
    * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically important history of liver disease, including viral or other hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with medical conditions that require the following medications will be excluded

  * Strong inhibitors of cytochrome P450 3A4 (CYP3A4) (clarithromycin, itraconazole, ketoconazole, nefazodone, erythromycin, grapefruit juice, verapamil, and diltiazem)
  * Strong inhibitors of cytochrome P450 2C9 (CYP2C9) (fluconazole and amiodarone)
  * Inducers of CYP3A4 (carbamazepine, dexamethasone, modafinil, oxcarbazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's wort, troglitazone)
  * Inducers of CYP2C9 (rifampin, and secobarbital)
* Patients who have a medical condition or dietary restrictions that prevent him or her from fasting for at least 10 hours (overnight) or eating a high calorie meal
* Any ambiguity in the inclusion/exclusion criteria should be clarified and resolved by communication with the study investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Vismodegib on Empty Stomach): Patients receive a single dose (150 mg) of vismodegib PO on an empty stomach. 7 days later, patients received 150 mg daily for 28 days.
  Pharmacological Study: Correlative studies
  Vismodegib: Given PO
- Arm II (Vismodegib After High Fat Meal): Patients receive a single dose (150 mg) of vismodegib PO after eating a high fat meal. 7 days later, patients received 150 mg daily for 28 days.
  Pharmacological Study: Correlative studies
  Vismodegib: Given PO
- Arm III (Vismodegib After Low Fat Meal): Patients receive a single dose (150 mg) of vismodegib PO after eating a low fat meal. 7 days later, patients received 150 mg daily for 28 days.
  Pharmacological Study: Correlative studies
  Vismodegib: Given PO
Period: Single Dose Pharmacokinetics
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Started | 23 | 20 | 20
Completed | 22 | 20 | 18
Not Completed | 1 | 0 | 2
Not completed — Early progressive disease | 1 | 0 | 1
Not completed — Patient entered hospice care | 0 | 0 | 1
Period: Steady-state Pharmacokinetics
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Started | 31 (Includes 22 patients from period 1 fasting arm and 9 patients from period 1 high-fat arm) | 0 (Patients in period 2 were randomized to fasting vs. fed state only.) | 29 (Includes 11 patients from period 1 high-fat arm and 18 patients from period 1 low-fat arm)
Completed | 25 | 0 | 27
Not Completed | 6 | 0 | 2
Not completed — Not evaluable | 6 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal) | Total
Number analyzed (Participants) | 23 | 20 | 20 | 63
Age, Continuous [Median (Full Range); unit: years] | 53 [34 to 74] | 57 [24 to 71] | 64 [46 to 84] | 61 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 14 | 40
  Male | 8 | 9 | 6 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 17 | 16 | 49
  African-American | 6 | 3 | 2 | 11
  Hispanic | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 20 | 20 | 63

OUTCOME MEASURES:

1. Primary Outcome: Cmax Following Single Dose of Drug
Description: Highest observed concentration over the 168 hour period. Blood samples were collected at j0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 24, 48, 120, and 168 hours.
Time Frame: 168 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 22 | 20 | 18
ng/ml | 3244 (55) | 5666 (45) | 3511 (40)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm II (Vismodegib After High Fat Meal); Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Performed on log-transformed data; Ratio of geometric means = 1.75, 90% CI 2-sided [1.30 to 2.34]
Statistical Analysis 2: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.65, t-test, 2 sided — Performed on log-transformed data; Ratio of geometric means = 1.08, 90% CI 2-sided [0.81 to 1.44]

2. Primary Outcome: AUC Following Single Dose of Drug
Description: Area under the curve from 0-168 hours.
Time Frame: 168 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 22 | 20 | 18
ng*h/mL | 416635 (56) | 723822 (54) | 466566 (38)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm II (Vismodegib After High Fat Meal); Test type: Superiority or Other; p = 0.008, t-test, 2 sided; Performed on log-transformed data; Ratio of geometric means = 1.74, 90% CI 2-sided [1.25 to 2.42]
Statistical Analysis 2: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.51, t-test, 2 sided; Performed on log-transformed data; Ratio of geometric means = 1.12, 90% CI 2-sided [0.84 to 1.49]

3. Secondary Outcome: Objective Responses in Patients With Solid Tumors
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 30 days
Population: 2 patients in Arm I and 4 patients in Arm III were non-evaluable for response.
Measure: Number; unit: participants
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 23 | 0 | 23
participants | 1 |  | 0

4. Primary Outcome: Tmax'Following Single Dose of Drug
Description: Time of maximum drug concentration
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 22 | 20 | 18
hours | 57 (62) | 44 (48) | 62 (57)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm II (Vismodegib After High Fat Meal); Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Tlag Following Single Dose of Drug
Description: Time between drug administration and when it is first observed in the systemic circulation.
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 22 | 20 | 18
hours | 0.11 (0.17) | 0.50 (0.29) | 0.58 (0.45)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm II (Vismodegib After High Fat Meal); Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Vismodegib on Empty Stomach); Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Ctrough Following Steady State Exposure for 14 Days
Description: Minimum blood concentration over 24-hour observation period. Blood sample collected at 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 24 hours.
Time Frame: 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 25 | 0 | 27
ng/ml | 10493 (37) |  | 12171 (35)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.17, t-test, 2 sided; Performed on log-transformed data; Ratio of geometric means = 1.16, 90% CI 2-sided [0.97 to 1.38]

7. Primary Outcome: Cmax Following Steady State Exposure for 14 Days
Description: Maximum drug concentration over 24 hours.
Time Frame: 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 25 | 0 | 27
ng/ml | 11449 (37) |  | 12950 (34)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.25, t-test, 2 sided; Performed on log-transformed data; Ratio of geometric means = 1.13, 90% CI 2-sided [0.95 to 1.35]

8. Primary Outcome: AUC Following Steady State Exposure for 14 Days
Description: Area under the curve from 0 to 24 hours.
Time Frame: 24 hours
Population: 3 and 2 patients with missing data, respectively
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 22 | 0 | 25
ng*h/mL | 238740 (40) |  | 290896 (35)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.096, t-test, 2 sided — Performed on log-transformed data; Ratio of geometric means = 1.22, 90% CI 2-sided [1.00 to 1.48]

9. Primary Outcome: Tmax Following Steady State Exposure for 14 Days
Description: Time of maximum drug concentration.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Number analyzed (Participants) | 25 | 0 | 27
hours | 6.7 (9.1) |  | 10.2 (10.3)
Statistical Analysis 1: Comparison: Arm I (Vismodegib on Empty Stomach) vs Arm III (Vismodegib After Low Fat Meal); Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: Includes all patients who received at least one dose in the daily dosing phase of the study. Recorded are adverse events of any grade level, whether or not attributable to the study drug.
Arm/Group | Arm I (Vismodegib on Empty Stomach) | Arm II (Vismodegib After High Fat Meal) | Arm III (Vismodegib After Low Fat Meal)
Serious Adverse Events (participants affected / at risk) | 15/31 | 0/0 | 14/30
Other Adverse Events (participants affected / at risk) | 31/31 | 0/0 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Vismodegib on Empty Stomach) (N=31) | Arm II (Vismodegib After High Fat Meal) (N=0) | Arm III (Vismodegib After Low Fat Meal) (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Death NOS (General disorders) | 5 | 0 | 3
Delirium (Psychiatric disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pain (General disorders) | 3 | 0 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Vismodegib on Empty Stomach) (N=31) | Arm II (Vismodegib After High Fat Meal) (N=0) | Arm III (Vismodegib After Low Fat Meal) (N=30)
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 5
Alanine aminotransferase increased (Investigations) | 4 | 0 | 8
Alkaline phosphatase increased (Investigations) | 9 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0 | 3
Anemia (Blood and lymphatic system disorders) | 14 | 0 | 10
Anorexia (Metabolism and nutrition disorders) | 15 | 0 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 6
Bloating (Gastrointestinal disorders) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 3 | 0 | 5
Chills (General disorders) | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 4 | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4
Creatinine increased (Investigations) | 4 | 0 | 3
Depression (Psychiatric disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 0 | 4
Dizziness (Nervous system disorders) | 4 | 0 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 8 | 0 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 8
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2
Edema limbs (General disorders) | 2 | 0 | 4
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fatigue (General disorders) | 13 | 0 | 15
Fever (General disorders) | 4 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Headache (Nervous system disorders) | 5 | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 0 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 0 | 5
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 0 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 5
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 6 | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 0 | 4
Hypotension (Vascular disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 0 | 1
Lymphocyte count decreased (Investigations) | 14 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 0 | 11
Non-cardiac chest pain (General disorders) | 3 | 0 | 3
Pain (General disorders) | 6 | 0 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 7
Platelet count decreased (Investigations) | 2 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 0 | 6
Weight loss (Investigations) | 7 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less